CLINICAL TRIAL: NCT04738721
Title: Comparison of Physical Activity and Physical Fitness Parameters Pre and Post COVID-19 Lockdown in Young Adults
Brief Title: Physical Activity and Physical Fitness Parameters in COVID-19 Lockdown
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, PhD, PT, Medipol University
Other Study IDs: E-10840098-772.02-2685
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Assessment, Self

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Evaluation — Within the scope of the course, the demographic information of the students (such as height, weight, body mass index) is recorded and the physical activity status is recorded with "International Physical Activity Questionnaire Short Form (UFAA)". Cardiovascular endurance with "6-Minute Walking Test", flexibility and circumference of waist, hip and neck with the "Sit and Lie Test" and body composition and "Body Fat Ratio "will be evaluated. After a full year of quarantine, the same students who were previously evaluated and accepted to participate in the current study will be evaluated with online remote video viewing methods (Teams, Zoom, etc.) and, with the same tests and measurements under supervision by the researchers.

SUMMARY:
In this study; it was aimed to compare the physical activity levels of students who continued their university education face-to-face before the COVID-19 lockdown, and the values of physical activity levels related to health, physical activity levels and health-related physical fitness parameters in the post-lockdown period.

DETAILED DESCRIPTION:
Within the scope of the course, the demographic information of the students will be recorded and physical activity status, physical fitness parameters, muscle endurance, cardiovascular endurance, flexibility and body composition will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Before the quarantine period, those who completed the physical activity level and physical fitness tests within the scope of Physical Activity I course
* Students who do not have any physical or mental problems for the tests and measurements to be applied

Exclusion Criteria:

* No internet access,
* Students who have an obstacle to taking tests and measurements

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of university
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Physical activity | 2 days
  International Physical Activity Questionnaire Short Form

SECONDARY OUTCOMES:
Physical fitness | 2 days
  6 Minute Walk Test
Flexibility | 2 days
  Sit-Rise Test
Body composition | 2 days
  Body fat ratio

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kaya Ciddi, PhD, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)